CLINICAL TRIAL: NCT02989818
Title: Multi-center Prospective Evaluation of the Clinical Utility of Endoscopic Submucosal Dissection (ESD) in the Western Population
Brief Title: Multi-center Evaluation of the Clinical Utility of ESD in the Western Population
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201600246
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Endoscopic Submucosal Dissection
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lesion of the Gastrointestinal tract: Investigator will collect prospective data on the Endoscopic Submucosal dissection that is used as part of the subjects standard of care to remove the Gastrointestinal lesion
  Interventions: Other: Endoscopic Submucosal Dissection

INTERVENTIONS:
Other: Endoscopic Submucosal Dissection — This intervention is part of the subjects standard of care and is a method to remove the Gastrointestinal lesion.
  Other Names: ESD

SUMMARY:
The aim of this multi-center study is to prospectively document the clinical utility of ESD.

DETAILED DESCRIPTION:
Multi-center prospective data recording study. All patients will receive standard medical care and no experimental interventions will be performed.

All patients scheduled to undergo ESD at the University of Florida and participating centers as medically indicated will be considered for the study. Patients in whom ESD is considered as part of their standard medical care will be offered to participate in this study. The physician performing the procedure will also discuss the study with the subjects. If the patient agrees to participate, he or she will be given the informed consent form and allowed enough time to read it. Opportunity to ask questions will be provided. If the patient agrees to participate, he or she will sign the consent form and a copy will be provided. Data will be prospectively recorded according to the data collection form. ESD will be performed as medically indicated. The investigators from each respective center on this project will also be in charge of the medical care of the patients enrolled in the study. Follow-up will be carried out as medically indicated and no additional studies or clinic visits will be needed specifically for the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* a. Age 18 years or older.
* b. Scheduled to undergo ESD as part of their standard of care.

Exclusion Criteria:

* a. Any contraindication to performing endoscopy.
* b. Participation in another research protocol that could interfere or influence the outcome measures of the present study.
* c. Patient is unable/unwilling to provide informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo ESD at the University of Florida and participating centers as medically indicated and part of their standard of care
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of en-bloc resection | 3-4 hours
  An Excision of the targeted lesion in a single specimen

SECONDARY OUTCOMES:
Rate of R0 resection | 3-4 hours
  when all vertical and horizontal margins are negative
Rate of R1 resection | 3-4 hours
  complete resection with no grossly visible lesion defined by endoscopist but microscopically positive horizontal and /or vertical margins
Curative resection | 3-4 hours
  this will have the following: R0 resection, Well to moderately differentiated histology, Absence of Lymphovascular invasion, Absence of budding, Absence of invasion beyond superficial submucosa
Rate of Adverse events with ESD | 1 month
  Early (<48 hours) and late (>48 hours) adverse events defined based on previously established criteria by the American Society of Gastrointestinal Endoscopy (ASGE)
Rate of complete remission of neoplasia | 1 month
  Absence of a visible lesion and/or absence of the neoplastic lesion on biopsy specimens (histopathology) obtained from the ESD site on follow up evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Peter Draganov, MD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] King W, Draganov P, Gorrepati VS, Hayat M, Aihara H, Karasik M, Ngamruengphong S, Aadam AA, Othman MO, Sharma N, Grimm IS, Rostom A, Elmunzer BJ, Yang D. Safety and feasibility of same-day discharge after endoscopic submucosal dissection: a Western multicenter prospective cohort study. Gastrointest Endosc. 2023 Jun;97(6):1045-1051. doi: 10.1016/j.gie.2023.01.042. Epub 2023 Jan 30. PMID 36731578
- [Derived] Yang D, King W, Aihara H, Karasik MS, Ngamruengphong S, Aadam AA, Othman MO, Sharma N, Grimm IS, Rostom A, Elmunzer BJ, Jawaid SA, Perbtani YB, Hoffman BJ, Akki AS, Schlachterman A, Coman RM, Wang AY, Draganov PV. Effect of endoscopic submucosal dissection on histologic diagnosis in Barrett's esophagus visible neoplasia. Gastrointest Endosc. 2022 Apr;95(4):626-633. doi: 10.1016/j.gie.2021.11.046. Epub 2021 Dec 11. PMID 34906544
- [Derived] Draganov PV, Aihara H, Karasik MS, Ngamruengphong S, Aadam AA, Othman MO, Sharma N, Grimm IS, Rostom A, Elmunzer BJ, Jawaid SA, Westerveld D, Perbtani YB, Hoffman BJ, Schlachterman A, Siegel A, Coman RM, Wang AY, Yang D. Endoscopic Submucosal Dissection in North America: A Large Prospective Multicenter Study. Gastroenterology. 2021 Jun;160(7):2317-2327.e2. doi: 10.1053/j.gastro.2021.02.036. Epub 2021 Feb 19. PMID 33610532